CLINICAL TRIAL: NCT00260715
Title: A Community-Based Intervention With Popular Opinion Leaders (C-POL) in Texas to Achieve Syphilis Elimination
Brief Title: A Community-Based Intervention With Popular Opinion Leaders (C-POL) in Texas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Texas A&M University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4133; U65/CCU622269; U65/CCU622268
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-12

CONDITIONS: Risk Behavior; Sexually Transmitted Diseases
Keywords: Risk behavior; Sexually Transmitted Diseases
MeSH Terms: conditions — Risk-Taking; Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Community-Popular Opinion Leader Model
Behavioral: Diffusion of Innovations

SUMMARY:
After exposure to the C-POL intervention: 1) unprotected vaginal or anal sex, sex with casual partners, concurrent sexual relationships, and exchange of sex for drugs or money will decrease significantly; 2) perceived syphilis-risk for self and peer group, knowledge about highly relevant risk-factors, information sources and resources will increase significantly; and 3) syphilis morbidity will decrease significantly in the intervention community as compared to the comparison community.

DETAILED DESCRIPTION:
The C-POL in Texas project is and intervention study which sought to impact the health behaviors of community residents who live in zip codes that have high syphilis morbidity. The study is being implemented in Texas (Dallas and Houston) with residents of a housing developing and the surrounding community.

The intervention model used for this study is the Popular Opinion Leader (POL) model, which is effective at reducing new HIV infections. The intent of this study was to determine the effectiveness of a diffusion model (e.g. POL) at reducing syphilis infections in affected communities.

For the intervention, community members identified as popular opinion leaders were recruited and trained to share accurate information about syphilis transmission, symptoms, testing, treatment and prevention. Prior to intervention implementation and several times after, community members were given a survey and screened for syphilis as well as 2-3 additional STDs. During each assessment, cross-sections of the community members were sampled.

ELIGIBILITY:
Inclusion Criteria:

* Community members who live and/or frequent the affected community. The affected community was one that had significant syphilis morbidity at the onset of the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2002-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Change in syphilis prevalence in affected community.

SECONDARY OUTCOMES:
Change in risk behaviors, and health care seeking.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Williams, Ph.D., Study Chair — CDC/NCHSTP/DSTDP/BIRB; Nilesh Chatterjee, Ph.D., Principal Investigator — Texas A&M University
Locations (1):
- Texas A& M University, College Station, Texas, United States